CLINICAL TRIAL: NCT05543538
Title: Influence of Different Teaching Strategies on the Academic Performance and Caring of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Taiwan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chiu Shu-Ching, assistant professor of nursing department, Central Taiwan University of Science and Technology
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: JAH.IRB.110-24
Record Dates: First submitted 2022-08-28; First posted 2022-09-16 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Nursing Students; Older People

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- multimedia audio-visual program (Placebo Comparator)
  Interventions: Other: multimedia audio-visual program
- multimedia audio-visual and experiential learning programmes (Experimental)
  Interventions: Other: multimedia audio-visual program; Other: experiential learning programmes
- multimedia audio-visual and teachers' personal demonstration and experiential learning (Experimental)
  Interventions: Other: multimedia audio-visual program; Other: experiential learning programmes; Other: teachers' personal demonstration

INTERVENTIONS:
Other: multimedia audio-visual program — Participants in the control group will receive teaching method with multimedia audio-visual material.
Other: experiential learning programmes — Participants in the experimental group will receive teaching method with experiential learning.
  Arms: multimedia audio-visual and experiential learning programmes; multimedia audio-visual and teachers' personal demonstration and experiential learning
Other: teachers' personal demonstration — Participants in the experience group will receive teachers' personal demonstration.
  Arms: multimedia audio-visual and teachers' personal demonstration and experiential learning

SUMMARY:
The participants in this study are college students with studying long-term care. After different teaching strategies, the students are hypothesised to improve their caring ability in the future and apply rhythmic muscle training programmes.

Therefore, this study will explore the relationship amongst three different teaching strategies of nursing students through multimedia audio-visual, multimedia audio-visual and experiential learning programmes and teachers' personal demonstration and experiential learning, as well as identify their relationship with caring ability.

ELIGIBILITY:
Inclusion Criteria:

1. Students aged 20 or above who have taken long-term care/long-term care-related courses.
2. Participate in this Community elders of the research project, aged 50 or above.

Exclusion Criteria:

1. No willingness to participate in the research.
2. Exercise taboos or physical health factors, such as severe frailty cases, severe illnesses Emotional instability, injury and inability to walk, pregnancy, etc.
3. Elders or students who cannot communicate in Chinese/Taiwanese.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Caring Assessment | 12 weeks
  5-Point Likert Scale and higher scores mean a better
Caring attitude | 12 weeks
  5-Point Likert Scale and higher scores mean a better
Caring Perception Behavior | 12 weeks
  5-Point Likert Scale and higher scores mean a better
Selfishness | 12 weeks
  2-point scales and higher scores mean more selfishness
behavioral intention of caring | 12 weeks
  5-Point Likert Scale and higher scores mean a better
The caring ability inventory | 12 weeks
  7-Point Likert Scale and higher scores mean a better
test for muscle strength training program | 12 weeks
  outcome for cognition aspect
idea transformation questionnaire | 12 weeks
  5-Point Likert Scale and higher scores mean a better
service-learning experience of scale for caring | 12 weeks
  6-Point Likert Scale and higher scores mean a better

SECONDARY OUTCOMES:
a caring scale for older adults | 12 week
  5-Point Likert Scale and higher scores mean a better

OTHER OUTCOMES:
Demographics | 12 weeks
  Religion, work, family interaction, activity related

CONTACTS AND LOCATIONS:
Overall Officials: Chiu, Principal Investigator — Central Taiwan University of Science and Technology
Locations (1):
- Central Taiwan University of Science and Technology, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No